CLINICAL TRIAL: NCT04692454
Title: Investigation of Immune Modulation by Modern Acupuncture in Gastroenterologic Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-Shun Wu, Director of GI, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N202005058
Record Dates: First submitted 2020-12-16; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Cancer; Gastrointestinal Cancer; Immunosuppression
Keywords: gastrointestinal; Hepatocellular; immunosuppression; acupuncture
MeSH Terms: conditions — Liver Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the scalp and ear acupuncture (Experimental): CHIAN HUEI ACUPUNCTURE NEEDLE
  Interventions: Other: Modern acupuncture

INTERVENTIONS:
Other: Modern acupuncture — use the scalp and ear acupuncture methods to identify diseases and checkpoints and apply them to regulate the immune function of patients with gastroenterological cancers.

SUMMARY:
According to the total population of cancer patients, hepatocellular carcinoma (HCC) and colorectal cancer (CRC), two of gastroenterological cancers are involved in the most acquired five cancers. Colorectal cancer (CRC) is a leading cause of tumor-related morbidity and mortality worldwide, and HCC is one of the top ten cancers in China. Currently, the intervention for gastrointestinal cancers mainly focuses on surgical removal, but patients still have a high risk of recurrence. Thus, the prevention of cancer recurrence is the most crucial topic for the intervention. The pathophysiology of gastroenterological cancers is multifactorial and not yet completely understood. However, immunosuppression is a major contributing factor in tumor cells play a central part in disease progression. It determines the prognosis of patients.

DETAILED DESCRIPTION:
According to the total population of cancer patients, hepatocellular carcinoma (HCC) and colorectal cancer (CRC), two of gastroenterological cancers are involved in the most acquired five cancers. Colorectal cancer (CRC) is a leading cause of tumor-related morbidity and mortality worldwide, and HCC is one of the top ten cancers in China. Currently, the intervention for gastrointestinal cancers mainly focuses on surgical removal, but patients still have a high risk of recurrence. Thus, the prevention of cancer recurrence is the most crucial topic for the intervention. The pathophysiology of gastroenterological cancers is multifactorial and not yet completely understood. However, immunosuppression is a major contributing factor in tumor cells play a central part in disease progression. It determines the prognosis of patients.

The immune checkpoint or complementary therapy in the course of cancer treatment has been reported as effective methods for patients. In recent years, more integrated treatment studies have found that acupuncture can improve the discomfort and pain caused by chemotherapy. In addition, the treatment of rheumatoid arthritis has shown that acupuncture can effectively regulate the immunity of patients. In this study, investigators are considering to apply modern acupuncture as the immune modulation in gastroenterological cancers. Modern acupuncture is to use the scalp and ear acupuncture methods to identify diseases and checkpoints and apply them to regulate the immune function of patients with gastroenterological cancers. The infiltration of a specific subtype of T-cell and the expression of PD-L1 in tumors may be applied as indicators of cancer prognosis. These CD8 T cells (also called Tex cells) often fail to eradicate tumors and can become dysfunctional or exhausted. The magnitude of the reinvigoration of circulating Tex cells determined in relation to pretreatment tumor burden correlated with clinical response. By monitoring Tex cells, investigators will evaluate the feasibility of acupuncture as a complementary therapy to regulate the immune functions of patients with gastroenterological cancers

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastrointestinal cancer
* Must have the will to receive acupuncture

Exclusion Criteria:

* Clinical diagnosis of Late cancer
* History of having bad reflect in acupuncture
* Coagulopathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The number of CD8+ T | 4 weeks
  Using PBMC to analyze the number of CD8+ T that is NK, NKT, DC, and Monocyte.
  At the start of acupuncture adjuvant therapy (week 0, week 2, and week 4) blood was collected.
  Blood draw - 15 ml/each
  Week0- baseline, the original data of CD8+T before receiving acupuncture
  Week2- the data of CD8+T after receiving acupuncture
  Week4- the data of CD8+T after two weeks that the patients did not receive acupuncture
  Compare with week0 and week2 data, if week2 data is higher than week0, it means the acupuncture has effective to add the number of CD8+ T.
  Compare with week 2 and week 4 data results and confirm the data change of the number of CD8+ T after stopping the acupuncture. If the data do not decline, it means the effect of acupuncture remains to exist. If the data declines, it means the effect of acupuncture weakens.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, PHD, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- WanFangH, Taipei, Taiwan